CLINICAL TRIAL: NCT05255237
Title: A Multicenter, Open-Label, Extension Study to Assess the Long-Term Safety and Efficacy of Jaktinib in Adult Patients With Moderate to Severe Alopecia Areata
Brief Title: Extension Study to Evaluate Safety and Efficacy of Jaktinib in Adults With Alopecia Areata
Acronym: AA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGJAK020
Record Dates: First submitted 2022-02-11; First posted 2022-02-24 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jaktinib (Experimental): Patients will administer the study product twice per day for 24 weeks, for the safety assessment.
  Interventions: Drug: Jaktinib

INTERVENTIONS:
Drug: Jaktinib — 75mg BID

SUMMARY:
This study (Unique Protocol ID: ZGJAK020) as an extension of the ongoing "Study to Evaluate Safety and Efficacy of Jaktinib in Adults With Alopecia Areata (Unique Protocol ID:ZGJAK020)" study. After completion of ZGJAK018 study, the study will be directly extend with an "open-label design".

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily sign the informed consent form.
* Patients who participated in ZGJAK018.

Exclusion Criteria:

* Subjects who are unsuitable to the trial, as identified by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting treatment-emergent adverse events | Baseline through week 24
  Patients with treatment-emergent adverse events/all patients *100%

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, PhD, Principal Investigator — Peking University People's Hospital; Qianjin Lu, PhD, Principal Investigator — Hospital for skin diseases, Chinese Academy of Medical Sciences
Locations (1):
- 11 Xizhimen South Street, Beijing, Beijing Municipality, China